CLINICAL TRIAL: NCT01361984
Title: Inspiratory Capacity and HRCT Comparison of Nebulized Arformoterol (Brovana) vs. Dry-powder Inhaler Salmeterol (Serevent)
Brief Title: Sunovion Brovana Versus Serevent Inspiratory Capacity High Resolution Computed Tomography
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Eric Kleerup, Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sunovion IC-HRCT
Record Dates: First submitted 2011-05-23; First posted 2011-05-27 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD; Emphysema; Chronic Bronchitis
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Emphysema; Chronic Bronchitis; Brovana; Serevent
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brovana (nebulized arformoterol) (Experimental): Brovana (nebulized arformoterol) treatment for 2 weeks
  Interventions: Drug: Nebulized arformoterol
- Serevent (Salmeterol dry powder inhaler) (Experimental): Serevent (Salmeterol dry powder inhaler) treatment for 2 weeks
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: Nebulized arformoterol — Arformoterol tartrate 15 µg/2ml (Brovana) nebulized via PARI-LC Plus® nebulizer with a mouthpiece, connected to a PRONEB® Ultra compressor. The nebulization time is ~9 minutes
  Other Names: Brovana
  Arms: Brovana (nebulized arformoterol)
Drug: Salmeterol — Salmeterol 50 mcg (Serevent) via Diskus dry powder inhaler
  Other Names: Serevent
  Arms: Serevent (Salmeterol dry powder inhaler)

SUMMARY:
This is a PI-initiated study taking place only at UCLA, sponsored by Sunovion. The investigators plan to enroll about 20 subjects who are at least 40 years old and have Chronic Obstructive Pulmonary Disease (COPD). The purpose of this study is to compare the effectiveness of Brovana and Serevent in helping relieve COPD symptoms. Specifically, the investigators are looking at how much and for how long the two drugs can open up the small airways in the lungs. This will be done with breathing tests on all subjects, and with high resolution CT scans on subjects who agree to this optional part of the study. Half of subjects will take Brovana (arformoterol tartrate inhalation solution) for 2 weeks and then Serevent (salmeterol xinafoate inhalation powder) for 2 weeks; the other half will take Serevent the first two weeks and Brovana the second two weeks. All subjects will also take Spiriva (tiotropium) and will be provided with albuterol for immediate relief of symptoms. After a Screening Visit to determine eligibility, subjects will be randomly assigned to receive Brovana or Serevent for the first 2 weeks, complete Test Visit 1, then receive the other study drug for 2 weeks, and finally complete Test Visit 2. Visits will include questionnaires, review of health and medications, and breathing tests before and after taking the study drug. Subjects who agree to be in the sub-study will also undergo CT scans before and after taking the study drug at both test visits.

ELIGIBILITY:
Inclusion Criteria:

* Age >=40 years
* History of smoking >=20 pack-years of cigarettes
* Be using medically acceptable birth-control measures if a female of child-bearing potential
* Be willing to withhold any existing short or long-acting bronchodilators for the appropriate time period prior to each test day. Use of inhaled corticosteroids is not exclusionary, but will be maintained at a constant level throughout the study.
* Must be willing and able to perform spirometry, slow vital capacity, plethysmography, DLCO, and 6 minute walk after appropriate instruction.
* Informed consent
* At the screening visit:

  * Post-albuterol FEV1/FVC <LLN (Hankinson)
  * Post-albuterol FEV1 <70%% and >=30 % predicted (Hankinson)
  * An increase in FEV1 after 4 puffs albuterol sulfate HFA of at least 5% and 50ml

Exclusion Criteria:

* Presence of other clinically significant illnesses or condition that might interfere with the study, including but not limited to uncontrolled hypertension, cardiovascular disease, cardiac arrhythmia, diabetes, hyperthyroidism, seizure disorder or any history of pheochromocytoma
* History of asthma (in the opinion of the investigator)
* A COPD exacerbations within the past 2 months requiring oral corticosteroids or hospitalization.
* Continuous oxygen therapy greater than 12 hours per day
* Subjects with a body mass index less than 15 or greater than 38
* Known allergy or contradiction to albuterol, arformoterol, salmeterol, tiotropium or prior significant adverse reactions to other beta agonists or ipratropium.
* Hypersensitivity to milk protein. Bloating or gas from lactose is not an exclusion.
* Inability to withhold other adrenergic drugs (salmeterol, arformoterol, formoterol, albuterol etc.) for an appropriate duration before each visit.
* Ongoing need for drugs which might potentiate hypokalemia (xanthine derivatives (theophylline), steroids, non-potassium sparing diuretics (unless in fixed combination with potassium sparing diuretic)
* Ongoing need for drugs which might cause QTc prolongation (MAO inhibitors, tricyclic antidepressants, cardiac anti-arrhythmics Class Ia (e.g., disopyramide, procainamide, quinidine), or class III (e.g., amiodarone, dofetilide, ibutilide, sotalol), terfenadine, astemizole, mizolastin and any other drug with potential to significantly prolong the QT interval.)
* Ongoing need for beta-blockers (selective or non-selective)
* Use of phenothizines (thioridizine), or other drugs that may interact with arformoterol, salmeterol or albuterol for the duration of the study. Washout of greater than seven half-lives of the drug prior to the study.
* History of angle closure glaucoma, symptomatic prostatic hypertrophy or bladder neck obstruction.
* Investigational drugs within 30 days
* Affiliation with the Division of Pulmonary and Critical Care Medicine, David Geffen School of Medicine
* Pregnancy, breastfeeding, planning to become pregnant during study, or woman of childbearing potential unwilling to use adequate contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Inspiratory capacity (absolute volume BTPS, L) | Week 4
  The inspiratory capacity (absolute volume BTPS, L) measured 3 times prior to treatment and 5-6 times after treatment will be contrasted between the two treatments (nebulized arformoterol and DPI salmeterol) using a mixed effects linear model. The model will include treatment order, albuterol response FEV1 in mL, time of day and whether the IC was from plethysmography and time of prior dose of study med (nominal 12 hours).

SECONDARY OUTCOMES:
Inspiratory capacity (absolute change, % change, %predicted change) | Week 4
  Inspiratory capacity: evaluated as absolute change, % change, %predicted change. Considered at predose (trough) and AUC 75-195 minutes after dose
Inspiratory capacity (%ref TLC) | Week 4
  Inspiratory capacity as percent of reference total lung capacity
Other breathing test outcomes | Week 4
  FEV1, FVC, isovolume FEF25-75% referenced to pre-albuterol FVC at screening visit, SVCexp (from spirometric and plethysmographic measures), FRC, RV, ERV, IRV, RV/TLC, TLC, IC/TLC

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States